CLINICAL TRIAL: NCT00007878
Title: A Phase I Study of PS-341 in Combination With 5-FU/LV in Solid Tumors
Brief Title: Bortezomib, Fluorouracil, and Leucovorin Calcium in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03190; NCI-2012-03190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-T99-0048; LAC-USC-0C003; CHNMC-PHI-27; CDR0000068327; PHI-27 (USC 0C-00-03) (Other: University of Southern California); T99-0048 (Other: CTEP); U01CA062505 (NIH)
Record Dates: First submitted 2001-01-06; First posted 2004-02-16 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bortezomib; Fluorouracil; Leucovorin

ARMS (1):
- Treatment (bortezomib, fluorouracil, leucovorin calcium) (Experimental): Patients receive bortezomib IV on days 1 and 4 and fluorouracil IV and leucovorin calcium IV on day 1 weekly for 2 weeks. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: fluorouracil; Drug: leucovorin calcium; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of bortezomib when given together with fluorouracil and leucovorin calcium in treating patients with solid tumors that are metastatic or cannot be removed by surgery. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with chemotherapy may be an effective treatment for solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of PS-341 (bortezomib) when administered as a bolus injection two times a week (on days 1 and 4) for 2 weeks followed by one week of rest.

II. To evaluate the pharmacodynamics of PS-341 by determining the 20S proteasome and nuclear factor kappa-light chain enhancer of activated B cells (NFkB) inhibition in blood of patients treated with intravenous PS-341 combined with weekly fluorouracil (5-FU) and leucovorin calcium (LV).

SECONDARY OBJECTIVES:

I. To identify any objective tumor response in patients treated with intravenous PS-341.

II. To evaluate the relationship between inhibition of the 20S proteasome and NFkB and clinical toxicity.

III. To obtain preliminary data on molecular correlates of response to PS-341 and 5-FU and LV including genes involved in apoptosis, cell cycle control, transcriptional regulation and adhesion/angiogenesis based on the mechanisms of PS-341 IV. To examine the pharmacokinetics of 5-FU when co-administered with PS-341.

OUTLINE: This is a dose-escalation study of bortezomib.

Patients receive bortezomib intravenously (IV) on days 1 and 4 and fluorouracil IV and leucovorin calcium IV on day 1 weekly for 2 weeks. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytological confirmed malignancy which is metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective
* All patients will have advanced malignancy confirmed by review of their biopsy specimens by the Division of Pathology of the City of Hope National Medical Center, the University of Southern California/LA County/Norris Comprehensive Cancer Center, or the University of California at Davis
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%) and an estimated survival of at least 3 months
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin =< within the institutional normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x the upper limits of institutional normal
* Serum creatinine =< 1.5 mg/dl
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, immunotherapy or radiotherapy within 4 weeks prior to entering the study and 6 weeks from nitrosourea-containing chemotherapy; all patients should have recovered from all toxicities of prior chemo and radiation therapy
* Patients undergoing therapy with other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other toxicities
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Pregnant and nursing women are excluded from this study because PS-341 is an investigational agent, and the anti-proliferative activity of PS-341 may be harmful to the developing fetus or nursing infant
* Human immunodeficiency virus HIV-positive patients receiving anti-retroviral therapy (HAART) are excluded from the study because of possible pharmacokinetic interactions
* Patients with electrocardiogram (EKG) evidence of acute ischemia or significant conduction abnormality (bifascicular block, defined as left anterior hemiblock in the presence of right bundle branch block, 2nd or 3rd degrees atrioventricular [AV] blocks); any history of cardiac or cerebrovascular disease due to hypotension and tachycardia
* Patients who had any major surgery within 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-09; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the highest dose tested in which none or only one patient experienced DLT attributable to the study drug(s), when at least 6 patients were treated at that dose and are evaluable for toxicity, graded according to the NCI CTC version 2.0 | Up to 21 days
Incidence of adverse events, graded according to NCI CTC version 2.0 | Up to 7 years
  The toxicities observed at each dose level will be summarized in terms of type, severity, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and course.

SECONDARY OUTCOMES:
Survival | Up to 7 years
  Will be summarized with Kaplan-Meier plots.
Time to failure | Up to 7 years
  Will be summarized with Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States